CLINICAL TRIAL: NCT07118462
Title: HighCycle Study: Effect of Acetazolamide on Plasma Volume During Acute Exposure to High Altitude in Women and Men
Brief Title: HighCycle Study: Acetazolamide, High Altitude and Plasma Volume
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre d'Expertise sur l'Altitude EXALT (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HighCycle_PV
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: High Altitude Effects; High Altitude Hypoxia; Acute Mountain Sickness (AMS); Plasma Volume; Women
Keywords: acetazolamide; plasma volume; acute mountain sickness; high altitude; hypoxia; women
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide 250 mg/day (capsules @125 mg; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules; 1 in the morning, 1 in the evening), orally. Medication starts 24 hours before ascent to 3600 m until the morning after the second night at 3600 m.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Administration of 1x125mg acetazolamide in the morning, 1x125mg in the evening, starting 24 hours before departure to 3600 m.
  Other Names: Diamox®
  Arms: Acetazolamide
Drug: Placebo — Administration of equally looking placebo capsules in the morning and in the evening, starting 24 hours before departure to 3600 m.
  Arms: Placebo

SUMMARY:
Each year, millions of people living at low altitude (< 1,000 m) travel to high altitude (≥ 2,500 m) for work, tourism, or sports activities. These individuals are exposed to hypobaric hypoxia, which can trigger acute mountain sickness (AMS)-the most common form of altitude-related illness. Therefore, understanding the physiological responses to hypoxia that allow acclimatization, as well as the pathophysiology of acute mountain sickness, is of primary importance.

The hematological response to high-altitude exposure initially includes a reduction in plasma volume (PV), leading to an early increase in hemoglobin concentration within the first 24 hours. In contrast, an increase in hemoglobin mass requires several weeks at high altitude. Recent well-controlled physiological studies conducted in hypobaric chambers have demonstrated that this hypoxia-induced PV contraction results from fluid redistribution from the intravascular to the extravascular compartment, rather than from water loss due to increased diuresis.

Prophylaxis of AMS is primarily based on the administration of 250 mg/day of acetazolamide (ACZ), a carbonic anhydrase inhibitor with a mild diuretic effect. Acetazolamide induces metabolic acidosis, which stimulates ventilation and thereby improves oxygenation. The effect of prophylactic ACZ use during high-altitude exposure on PV in lowlanders remains unknown: it is unclear whether ACZ leads to a greater reduction in PV due to its diuretic effect, or to a smaller hypoxia-induced PV contraction as a result of improved oxygenation induced by increased ventilation.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking men and women, age 18-44 years, without any disease and need of regular medication (including oral contraceptives).
* BMI >18 kg/m2 and <30 kg/m2.
* Born, raised and currently living at altitudes <1000 m.
* Written informed consent.
* Premenopausal women with an eumenorrheic cycle.

Exclusion Criteria:

* Other types of contraceptvies (contraceptives (hormonal intrauterine device, vaginal ring, subcutaneous injections or implants, among others).
* Pregnancy or nursing
* Anaemic (haemoglobin concentration <10g/dl).
* Any altitude trip <4 weks before the study.
* Allergy to acetazolamide and other sulfonamides.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma volume | Day 1 at 760 m then Day 2 and Day 3 at 3,600 m.
  Change in plasma volume assessed by the CO-rebreathing method in acetazolamide versus placebo group

SECONDARY OUTCOMES:
Plasma volume : sex-related difference | Day 1 at 760 m then Day 2 and Day 3 at 3600 m.
  Sex-related differences in the effect of acetazolamide vs.placebo in plasma volume at high altitude.
Plasma volume : AMS-related difference | Day 1 at 760 m then Day 2 and Day 3 at 3600 m.
  Difference in plasma volume change at high altitude between AMS+ and AMS- participants.
Hormones | Day 2 at 760 m and Day 2 at 3600 m.
  Changes in copeptin and midregional proANP serum levels between acetazolamide and placebo group and sex-related difference
Arterial blood gases | Day 2 at 760 m and Day 2 at 3600 m.
  Changes in the arterial blood gases (pH, PaO2, PaCO2, SaO2) between acetazolamide and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furian, Prof. Dr., Study Chair — University of Zurich; Talant M Sooronbaev, Prof. Dr., Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Paul Robach, PhD, Principal Investigator — EXALT (Centre d'Expertise sur l'Altitude), Grenoble, France; Benoit Champigneulle, MD, PhD, Principal Investigator — EXALT (Centre d'Expertise sur l'Altitude), Grenoble, France
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication